CLINICAL TRIAL: NCT02781194
Title: A Prospective, Randomized, Controlled, Study Investigating Intraoperative Temperature and Postoperative Pain Course Following Gynaecological Laparoscopy
Brief Title: Temperature and Pain in Laparoscopy
Acronym: TePaLa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 13-030
Record Dates: First submitted 2016-05-17; First posted 2016-05-24 (Estimated); Last update posted 2019-02-12 (Actual); Status verified 2018-02

CONDITIONS: Intraoperative Temperature; Postoperative Pain; Laparoscopy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- forced-air warming blanket (Experimental): Forced-air warming blanket via 3M™ Bair Hugger™.
  Interventions: Device: 3M™ Bair Hugger™
- warmed, humidified insufflation (Experimental): Warmed, humidified insufflation via the F&P HumiGard™ Surgical Humidification System.
  Interventions: Device: F&P HumiGard™ Surgical Humidification System
- forced-air warming blanket & warmed, humidified insufflation (Experimental): Combination of forced-air warming blanket via 3M™ Bair Hugger™ and warmed, humidified insufflation via the F&P HumiGard™ Surgical Humidification System.
  Interventions: Device: 3M™ Bair Hugger™; Device: F&P HumiGard™ Surgical Humidification System

INTERVENTIONS:
Device: 3M™ Bair Hugger™ — forced-air warming blanket
  Arms: forced-air warming blanket; forced-air warming blanket & warmed, humidified insufflation
Device: F&P HumiGard™ Surgical Humidification System — warmed, humidified insufflation
  Arms: forced-air warming blanket & warmed, humidified insufflation; warmed, humidified insufflation

SUMMARY:
The aim of this investigation is to assess the impact of forced air warming, warm humidified insufflation gas and the combination of the two on intraoperative temperature maintenance and the postoperative pain course as well as the fibrinolytic activity in peritoneal fluid following laparoscopic procedures (duration > 60 min) in a prospective, randomized, controlled, mono-centric study. Therefore 150 subjects will be randomized in 3 groups of 50 subjects each. First group will be treated with forced-air warming blanket (bair hugger). Second group will be treated with warmed, humidified insufflation via the F&P HumiGard™ Surgical Humidification System. Third group will be treated with both, warming blankets and warmed, humidified insufflation. The peri-operative temperature of patients might be higher in patients of the third group with the combination of both treatments. The investigators hypothesize that VAS scores for pain (especially shoulder pain), and MEDD usage will differ between groups. Wound infection incidence and time spent in PACU are also expected to differ. Fibrinolytic activity in the peritoneal fluid is expected to be higher in patients undergoing laparoscopic procedures with humidified gas insufflation, since the trauma to the peritoneum will be less.

DETAILED DESCRIPTION:
During the first 30 to 40 minutes of anaesthesia, a patient's temperature can drop to below 35.0°C. Reasons for this include loss of the behavioural response to cold and the impairment of thermoregulatory heat-preserving mechanisms under general or regional anaesthesia, anaesthesia-induced peripheral vasodilation, the use of cold dry insufflation gases. For these reasons, institutions employ a range of techniques to prevent hypothermia, including forced air warming (peri-operatively), use of warmed intravenous fluids, temperature monitoring and control of room temperature. Despite these interventions audits demonstrate that 20-56% of patients are hypothermic during the perioperative period. A factor often dismissed as a cause of peri-operative hypothermia during laparoscopic procedures is dry and cold insufflation gas. During laparoscopic procedures the abdomen is continuously insufflated with cold, dry CO2 resulting in desiccation and heat loss which consequently induces hypothermia in the patient. Clinical evidence suggests that the risk of hypothermia can be reduced using warm and humidified gas, as has been shown in animal models, in clinical trials and confirmed in a metaanalysis in humans. Only gas at body temperature and fully saturated with moisture will prevent loss of energy from the peritoneum surface - because it is physically not possible to evaporate fluids into a fully saturated gas. Therefore, the fluid layer will be maintained, minimizing energy loss from the body, decreasing the hypothermia induced by the evaporative losses in laparoscopic surgery and stabilizing the fibrinolytic activity of the peritoneum. The aim of this investigation is to assess the impact of forced air warming, warm humidified insufflation gas and the combination of the two on intraoperative temperature maintenance and the postoperative pain course as well as the fibrinolytic activity in peritoneal fluid following laparoscopic procedures (duration > 60 min) in a prospective, randomized, controlled, mono-centric study. Therefore 150 subjects will be randomized in 3 groups of 50 subjects each. First group will be treated with forced-air warming blanket (bair hugger). Second group will be treated with warmed, humidified insufflation via the F&P HumiGard™ Surgical Humidification System. Third group will be treated with both, warming blankets and warmed, humidified insufflation. The peri-operative temperature of patients might be higher in patients of the third group with the combination of both treatments. The investigators hypothesize that VAS scores for pain (especially shoulder pain), and MEDD usage will differ between groups. Wound infection incidence and time spent in PACU are also expected to differ. Fibrinolytic activity in the peritoneal fluid is expected to be higher in patients undergoing laparoscopic procedures with humidified gas insufflation, since the trauma to the peritoneum will be less.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or above and aged under 70 years
* Written informed consent prior to study participation
* Patients admitted to hospital for laparoscopic surgery with a planned duration of more than 1 hour; if there is an open component to the surgery then this should be discussed, in terms of the length of the laparoscopic component
* BMI <35

Exclusion Criteria:

* Pregnancy or women without sufficient contraception
* Women, who are breastfeeding
* Alcohol or drug abuse
* Expected non-compliance
* Patients unwilling or unable to give informed consent, patients with limited ability to comply with instructions for this study
* Participation on another interventional study within the last 3 months
* Subjects who are committed to an institution and/or penitentiary by judicial or official order
* Employees of the investigator cooperation companies

Ages: 18 Years to 69 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Intra-operative core temperature | 2 hours
  Intra-operative core temperature measured via oesophageal probe/urinary catheter after anaesthetic induction (baseline) but before insufflation and at 10 minute intervals until completion of surgery; hypothermia (<36 C) during the peri-operative period to be indicated by:
  * Mild (core temperature 35.0 °C to 35.9 °C)
  * Moderate (34.0 °C to 34.9 °C)
  * Severe ≤33.9 °C)
Body temperature | 2 hours
  Body temperature as measured by direct tympanic thermometer:
  * Pre-operatively - 1 hour before induction and at 10 minute intervals until induction
  * Before anesthetic induction
  * Post-operatively at entry to recovery room and at 10 minute intervals or until normo-thermia (≥36.5 °c) is achieved. Time at which normothermia is achieved to be recorded.
VAS (visual analouge scale): composite measure of pain in different regions of the body | up to 7 days
  VAS: Pain from abdominal area - Pain in the shoulder
  - Pain on movement - Pain on coughing, before transfer to ward; at arrival in recovery room; 8 a.m. + 8 p.m. until discharge; 0 - 10 Numeric Pain Rating Scale by VAS, National Institute of Pain Control - NIPCTM
morphine equivalent daily dose (MEDD) usage in patient controlled analgesia (PCA) | up to 7 days
  MEDD usage: intraoperative, post anaesthesia care unit (PACU), Day 0, Day 1, Day 2, Day 3, Total during admission, Day on which PCA is removed if PCA is used. Start of PCA to be standardised, if possible all patient requests for PCA to be recorded by software, even if patient lockout has occurred due to too many attempts to activate PCA in a certain time.
Perioperative Fluid (PV) | 2 hours
  PV to be recorded at 10 min intervals perioperatively. Volume of electrolyte solution infused to be recorded, as well as time from induction until infusion takes place.
Fibrinolytic activity | 2 days
  Fibrinolytic activity in the peritoneal fluid will be determined at the beginning of surgery and Day 1. Sample will be taken from an abdominal drain.

CONTACTS AND LOCATIONS:
Overall Officials: Julia Wittenborn, Dr. med., Principal Investigator — Uniklink RWTH Aachen, Klinik für Gynäkologie und Geburtsmedizin
Locations (1):
- Uniklink RWTH Aachen, Klinik für Gynäkologie und Geburtsmedizin, Aachen, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] 1. Frank S, Fleisher L, Breslow M, et al. Perioperative maintenance of normothermia reduces the incidence of morbid cardiac events. A randomized clinical trial [see comments]. JAMA 1997; 277(14):1127-34. -- 2. Frank S, Higgins M, Fleisher L, et al. Adrenergic, respiratory, and cardiovascular effects of core cooling in humans. Am J Physiol 1997; 272(2 Pt 2):R557-62. -- 3. Kurz A, Sessler DI, Lenhardt R. Perioperative normothermia to reduce the incidence of surgical-wound infection and shorten hospitalization. New England Journal of Medicine 1996; 334(19):1209-1215. -- 4. Hofer CK, Worn M, Tavakoli R, et al. Influence of body core temperature on blood loss and transfusion requirements during off-pump coronary artery bypass grafting: a comparison of 3 warming systems. J Thorac Cardiovasc Surg 2005; 129(4):838-43. -- 5. Johansson T, Lisander B, Ivarsson I. Mild hypothermia does not increase blood loss during total hip arthroplasty. Acta Anaesthesiol Scand 1999; 43(10):1005-10. -- 6. Melling AC, Ali B, Scott EM, Leaper DJ. Effects of preoperative warming on the incidence of wound infection after clean surgery: a randomised controlled trial.[see comment][erratum appears in Lancet 2002 Mar 9;359(9309):896]. Lancet 2001; 358(9285):876-80. -- 7. Nesher N, Zisman E, Wolf T, et al. Strict thermoregulation attenuates myocardial injury during coronary artery bypass graft surgery as reflected by reduced levels of cardiac-specific troponin I. Anesth Analg 2003; 96(2):328-35, table of contents. -- 8. Persson K, Lundberg J. Perioperative hypothermia and postoperative opioid requirements. Eur J Anaesthesiol 2001; 18(10):679-86. -- 9. Schmied H, Kurz A, Sessler DI, et al. Mild hypothermia increases blood loss and transfusion requirements during total hip arthroplasty. Lancet 1996; 347(8997):289-92. -- 10. Sellden E. Peri-operative amino acid administration and the metabolic response to surgery. Proc Nutr Soc 2002; 61(3):337-43.
- [Derived] Wittenborn J, Mathei D, van Waesberghe J, Zeppernick F, Zeppernick M, Tchaikovski S, Kowark A, Breuer M, Keszei A, Stickeler E, Zoremba N, Rossaint R, Bruells C, Meinhold-Heerlein I. The effect of warm and humidified gas insufflation in gynecological laparoscopy on maintenance of body temperature: a prospective randomized controlled multi-arm trial. Arch Gynecol Obstet. 2022 Sep;306(3):753-767. doi: 10.1007/s00404-022-06499-z. Epub 2022 Mar 14. PMID 35286431
- [Derived] Breuer M, Wittenborn J, Rossaint R, Van Waesberghe J, Kowark A, Mathei D, Keszei A, Tchaikovski S, Zeppernick M, Zeppernick F, Stickeler E, Zoremba N, Meinhold-Heerlein I, Bruells C. Warm and humidified insufflation gas during gynecologic laparoscopic surgery reduces postoperative pain in predisposed patients-a randomized, controlled multi-arm trial. Surg Endosc. 2022 Jun;36(6):4154-4170. doi: 10.1007/s00464-021-08742-1. Epub 2021 Oct 1. PMID 34596747